CLINICAL TRIAL: NCT01418924
Title: Effects Of Sex Hormones On Serum Sclerostin Level During Menstrual Cycle
Brief Title: Sex Hormones & Serum Sclerostin Level
Acronym: SHSCL
Status: Completed | Type: Observational
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Karacan, Chief of Physical Med & Rehab Clinic, Bagcilar Training and Research Hospital
Other Study IDs: BEAH FTR-4
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Bony Sclerosis; Testicular; Hormone, C
Keywords: sclerostin; estradiol; progesterone; testosteron; sex hormones
MeSH Terms: conditions — Sclerosteosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to determine whether plasma sclerostin levels is affected by sex hormones during menstrual cycle. Blood samples will be obtained at the beginning (between 2-5th day), mid (between 11-13th day) and end (between 21-23th day) of menstrual cycle. Serum sclerostin, estradiol, progesterone and testosteron levels will be measured blindly by only one investigator

DETAILED DESCRIPTION:
This study is a prospective, observational, single-center study. Ethical approval was obtained from the Institutional Review Board.

This study will be completed with 40 premenopausal healthy volunteer women. An intravenous cannula will be inserted into the antecubital vein. Blood samples will be obtained at the beginning (between 2-5th day), mid (between 11-13th day) and end (between 21-23th day) of menstrual cycle.

Serum will be collected and will be centrifuged for 15 minutes at 1000Xg within 30 minutes of collection. Aliquots of plasma will be added to Ependorf tubes and stored at -20°C.

Plasma sclerostin levels will be measured using a Human Sclerostin ELISA kit (Cusabio, Catalog No: CSB-E13146h, Newark, DE, USA). All assays will be performed according to the manufacturer's instructions. The minimum detectable concentration of human sclerostin is typically <0.012 ng/ml. Intra-assay precision is less than 8%.

Estradiol and progesterone levels will be analyzed in serum samples using an electrochemiluminescence immunoassay (Elecsys PTH, Elecsys-estradiol II; Roche Diagnostics, Mannheim, Germany) and the Cobas 601 analyzing system (Roche Diagnostics).

Free testosteron levels will be analyzed in serum samples using an RIA (radio immun assay) (DSL 4900 Testosterone, Free, Active® RIA Assay kit, Beckman Coulter) and the DSL 4900 Berthold Technologies Multi Crystal LB 2111 model gama counter.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal women
* healthy
* volunteer

Exclusion Criteria:

* Endocrinopathies
* Bone disease (osteoporosis, osteomalacia, paget disease etc)
* Women who used hormonal drug within last six months
* Cognitive disorders

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Premenopausal healthy women
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Serum sclerostin level | 1 month
  Changes in serum sclerostin level by sex hormons during menstrual cycle

CONTACTS AND LOCATIONS:
Overall Officials: MUHARREM CIDEM, MD, Principal Investigator — Bagcilar Training & Research Hospital Istanbul, Turkey
Locations (1):
- Bagcilar Training & Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Cidem M, Usta TA, Karacan I, Kucuk SH, Uludag M, Gun K. Effects of sex steroids on serum sclerostin levels during the menstrual cycle. Gynecol Obstet Invest. 2013;75(3):179-84. doi: 10.1159/000347013. Epub 2013 Feb 21. PMID 23429230